CLINICAL TRIAL: NCT05306951
Title: Correct Timing of Head Imaging in Trauma
Acronym: CT-HIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Padova (Other)
Collaborators: University Hospital Padova (Other)
Responsible Party: Principal Investigator, Giulia Berti de Marinis, Principal investigator, University Hospital Padova
Other Study IDs: PDED0121
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Craniocerebral Trauma; Platelet Aggregation Inhibitors
MeSH Terms: conditions — Craniocerebral Trauma | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Computed tomography — Head computed tomography
  Other Names: Single computed tomography

SUMMARY:
The aims of this retrospective and monocentric observational study are: to describe patient characteristics and clinical management of patients with traumatic brain injury taking antiplatelet and/or anticoagulation drugs; to estimate the proportion of patients who suffer an adverse outcome; to assess the risk for serious events (intracranial haemorrhage, in-hospital mortality, need for surgery); to identify potential predictors of outcome and assess potential differences between anticoagulation and antiplatelet therapy.

All patients with mild brain injury and anticoagulant or antiplatelet therapy who underwent a head computed tomography (CT) scan admitted to the emergency department (ED) of the University Hospital of Padova, Italy, from 01/01/2010 to 31/12/2020.

DETAILED DESCRIPTION:
Background Mild traumatic brain injury (mTBI) is one of the most common occurrences at the emergency departments in Italy and worldwide constituting major health and socioeconomic issue all over the world. mTBI is defined as a patient reporting a Glasgow Coma Scale (GSC) score of 14-15, disorientation, amnesia and loss of consciousness. On the other hand, the patient population treated with anticoagulant or antiplatelet drug therapy is increasing: this therapy is prescribed to prevent thromboembolic complications of atrial fibrillation, deep venous thrombosis, and surgically placed cardiac valves, especially in the elderly population. Numerous studies suggested that mostly aged patients or those with comorbidities with mTBI on anticoagulant or antiplatelet drug therapy have a higher risk of developing a haemorrhagic complication; but there is a lack of evidence for patients on new anticoagulants and second-generation antiplatelet drugs regarding a higher risk for intracranial haemorrhage (ICH), ICH progression, or death. Several international guidelines have been developed for the management of traumatic brain injury and they all recommended performing brain computed tomography (CT) for patients with head trauma taking oral anticoagulant agents even in absence of any neurological symptoms. Nevertheless, there is no agreement about the correct timing for performing a head CT scan, the duration of observation before discharge from ED and the necessity of repeating a second CT scan at distance. National Institute for Health and Care Excellence (NICE) guidelines 2014 recommend performing a CT scan within 8 hours of the injury for patients on anticoagulant therapy with mTBI and no other neurological symptoms, while European Federation of the Neurological Societies (EFNS) guidelines 2008 and New South Wales (NSW) guidelines 2011 recommend observation for 24 h and considering a second CT scan. A recent meta-analysis has collected 24 significant studies investigating the incidence of delayed intracranial haemorrhage in patients presenting with mTBI and anticoagulant or antiplatelet drug therapy: as far as anticoagulant drug therapy is concerned, only 2 studies regarding patients on double oral anticoagulation (DOAC) and 14 studies regarding patients on Vitamine K Antagonists (VKA) were identified. The incidence of delayed intracranial haemorrhage in both groups was the same (1.3%) and no difference was found between patients on DOAC who underwent a single CT scan and a repeated one after observation.

Main objective To describe patient characteristics and clinical management of patients with a head injury during antithrombotic therapy To assess the risk for serious events (intracranial haemorrhage, death for traumatic brain injury, need for surgery) in patients on anticoagulant therapy and/or antiplatelet drugs who underwent a head CT scan following head injury.

To identify potential predictors of outcome and assess potential differences between anticoagulation and antiplatelet therapy.

Study design Retrospective, single centre non-interventional study of all patients admitted to the emergency department (ED) of the University Hospital of Padova, Italy, from 01/01/2010 to 31/12/2020, for traumatic brain injury. All patients on anticoagulant therapy and antiplatelet drugs who underwent a head CT scan will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* A head computed tomography (CT) scan following head trauma
* Age ≥18 Years
* Anticoagulant and/or antiplatelet therapy

Exclusion Criteria:

* moderate or severe brain injury (GCS ≤ 13 in the initial assessment in the ED)
* concomitant severe thoracic trauma with hypoxia (satO2 < 90% room air)
* active bleeding and/or hemodynamic instability
* intracranial haemorrhage with features suggesting spontaneous bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mild brain injury and anticoagulant or antiplatelet therapy who underwent a head CT scan and have been admitted to the Emergency Department
Sampling Method: Non-Probability Sample
Enrollment: 3200 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of intracranial hemorrhage | 30 days
  Diagnosis of intracranial hemorrhage

SECONDARY OUTCOMES:
Need for surgery at 30-days-follow-up | 30 days
  Need for surgery at 30-days-follow-up
Mortality for traumatic brain injury at 30-days-follow up | 30 days
  Mortality for traumatic brain injury at 30-days-follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedale Università Padova, Padua, PD, Italy

IPD SHARING:
Plan to Share IPD: Undecided